CLINICAL TRIAL: NCT03188354
Title: Diagnostic Assessment of 18F-fluciclovine and 18F-FDG - PET/MRI of Primary Central Nervous System Lymphoma
Brief Title: Diagnostic Assessment of 18F-fluciclovine and 18F-FDG -PET/MRI of Primary Central Nervous System Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET/MRI_CNS_LYMPHOMA; 2017-000306-38 (EudraCT Number)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma, Non-Hodgkin; Central Nervous System Neoplasms
Keywords: Positron-Emission Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Central Nervous System Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNS lymphoma patients (Experimental): Patients included in the study will be examined with both 18F-FDG and 18F-Fluciclovine as well as standard MRI in the PET/MRI scanner on two consecutive days, both in primary staging and for therapy assessment
  Interventions: Diagnostic Test: 18F-FDG; Diagnostic Test: 18F-fluciclovine; Diagnostic Test: standard MRI

INTERVENTIONS:
Diagnostic Test: 18F-FDG — PET scan with 18F-FDG as a tracer, taken both for primary staging and therapy assessment.
  Other Names: Fluorine-18 Fluorodeoxyglucose
Diagnostic Test: 18F-fluciclovine — PET scan with 18F-fluciclovine as a tracer, taken both for primary staging and response to therapy assessment.
  Other Names: amino-acid PET-tracer
Diagnostic Test: standard MRI — clinical routine MRI examination, both for primary staging and response to therapy assessment.
  Other Names: Magnetic resonance imaging

SUMMARY:
Primary central nervous system lymphoma (PCNSL) is a rare subtype of extranodal non-Hodgkins Lymphoma (NHL) with rising incidence and variable response to treatment. MRI is considered the most useful imaging modality of PCNSL, but conventional MRI has its limitations, and contrast-enhanced MRI sometimes does not clearly differentiate PCNSL from other neoplasm or non-neoplastic diseases.

Positron emission tomography (PET) could have a number of potential advantages in refining and improving the management of patients with PCNSL. Because of the rare incidence of PCNSL, the value of PET has however not been well defined in this subtype of lymphomas. There are a few studies that have investigated the role for FDG-PET and amino acid PET in the primary staging/diagnosis and response assessment in PCNSL patients, but the results are inconclusive. Further studies are therefore needed.

Previous studies support an integration of both MRI and PET for the routine diagnostic workup and response assessment for PCNSL, and the newly available simultaneous PET/MRI scanners may have the potential to improve imaging baseline accuracy, response assessment and add prognostic value in PCNSL.

The main aim of the study is to compare the sensitivity and specificity of a combined PET/MRI examination with the clinical routine MRI examination given to these patients today. It will be investigated whether PET (18F-FDG and 18F-fluciclovine) can provide additional prognostic value at baseline and in response assessment compared to MRI and established pre-treatment prognostic scores in PCNSL, and evaluate which PET/MRI parameters that are best suited as an imaging biomarker for progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of PCNSL based on cytology/flow cytometry of cerebrospinal fluid (CSF) or brain biopsy
* Written informed consent from patient or guardian
* Immunocompetent

Exclusion Criteria:

* Previous chemotherapy
* Contra-indications for MRI (Pacemakers, defibrillators, aneurysm clips, any form of metal in the body, or severe claustrophobia)
* Hypersensitivity to either 18F-Fluciclovine or 18F-FDG or to any of the excipients
* Pregnancy (pregnancy test for all women in fertile age)
* Breastfeeding
* Weight > 120 kg
* Estimated glomerular filtration rate (eGFR) <30ml/min/1,73m2
* HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of 18F-Fluciclovine-PET/MRI sans | 2 days
  of combined 18F-Fluciclovine-PET/MRI examination in comparison with the clinical routing MRI examination
sensitivity and specificity of 18F-FDG-PET/MRI scans | 2 days
  of combined 18F-FDG-PET/MRI examination in comparison with the clinical routing MRI examination

SECONDARY OUTCOMES:
prediction of progression-free survival | 1 year
  which PET/MRI parameters that are best suited as an imaging biomarker for response evaluation and for progression-free survival at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, phd, Study Director — Norwegian University of Science and Technology, Department of Circulation and Medical Imaging
Locations (1):
- Norwegian University of Science and Technology, Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Husby T, Johannessen K, Berntsen EM, Johansen H, Giskeodegard GF, Karlberg A, Fagerli UM, Eikenes L. 18F-FACBC and 18F-FDG PET/MRI in the evaluation of 3 patients with primary central nervous system lymphoma: a pilot study. EJNMMI Rep. 2024 Jan 31;8(1):2. doi: 10.1186/s41824-024-00189-6. PMID 38748286